CLINICAL TRIAL: NCT06632158
Title: Personal Relevance of Psychotherapy for Asian Americans: A mHealth Problem-solving Intervention to Reduce Stress (PRoP-AA)
Brief Title: Personal Relevance of Psychotherapy for Asian Americans
Acronym: PRoP-AA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRIS Media Inc (Other)
Responsible Party: Principal Investigator, Jordan Pennefather, Senior Scientist, IRIS Media Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4R44MH125698-02 (NIH)
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Behavior; Stress; Anxiety
Keywords: Problem-Solving Therapy; Online App; MindBoba
MeSH Terms: conditions — Behavior; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Three-arm design comparing the new intervention (MindBoba) to an active control (Mindshift CBT) and business-as-usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MindBoba (Experimental): Participants will be given access to the MindBoba app for 12 weeks.
  Interventions: Behavioral: MindBoba
- Mindshift CBT (Active Comparator): Participants will be given access to the Mindshift CBT app for 12 weeks.
  Interventions: Behavioral: Mindshift CBT
- Business-as-Usual (No Intervention)

INTERVENTIONS:
Behavioral: MindBoba — MindBoba is a smartphone app that uses strategies based on Problem-Solving Therapy to help decrease stress and anxiety, and teach new skills.
  Arms: MindBoba
Behavioral: Mindshift CBT — MindShift® CBT uses strategies based on Cognitive Behavioural Therapy (CBT) to help participants learn to relax and be mindful, develop more effective ways of thinking, and use active steps to take charge of their anxiety.
  Arms: Mindshift CBT

SUMMARY:
Using a three-armed design the investigators will test whether participants in the Mindboba online application experience significantly greater improvements as compared to participants in the active control (online app based on Cognitive Behavioral Therapy) and participants in the business-as-usual control. The outcome measures are self-reported social problem-solving, self-efficacy, stress, depression, anxiety, attitudes towards seeking mental health, and knowledge.

DETAILED DESCRIPTION:
The intervention, Personal relevance of psychotherapy for Asian Americans: A mHealth problem-solving intervention to reduce stress, is designed 1) to increase the use of mental health services by a population that uses them at one third the rate of Whites,and 2) to develop a personally-relevant approach to stress-reduction. Practical and cultural barriers inhibit the use of mental health services by Asian Americans including a lack of fluency in English amongst specific subpopulations, insufficient health literacy, and stigma surrounding mental illness which stems from Asian American cultural beliefs shared across subpopulations. To this end the investigators developed MindBoba a mHealth (mobile health) application that is systematically adapted to be culturally relevant to select Asian American subpopulations based on Problem-Solving Therapy (PST).

To ensure client engagement, psychotherapy should provide relevant, immediate, and tangible benefits. Personally relevant, evidence-based interventions have the potential to increase the reach and impact of mental health services-especially as conventional, evidence-based interventions have not worked to eliminate mental health disparities among ethnic minority groups. Personally relevant interventions can reduce disparities by increasing engagement, and greater engagement makes mental health services more effective. An external problem-solving orientation is culturally responsive to Asian values. It focuses on the problem, allowing the client to feel more comfortable in treatment, rather than on cognitive reframing, which can elicit an aversive reaction if the client is unprepared to make internal shifts and feels blamed when asked by the therapist to do so. By approaching personal issues as external problems to solve, as opposed to a personal disease to manage, Asian Americans can effectively save face, a particular concern. PST is effective for reducing psychopathology, such as depression and other psychological difficulties. Research has shown that Asian Americans report greater perceived relevance of PST, as well as greater activation of self-processing, in the medial prefrontal cortex compared to Cognitive Behavioral Therapy (CBT).

The MindBoba intervention's content is innovative, it integrates external problem-solving and goal-setting through the use of PST. By focusing on stressful problems in the real world, PST offers a more personally relevant approach for many Asian Americans-particularly those concerned about saving face. Mindboba was culturally adapted for this group systematically. Culturally adapted strategies may include providing cultural-clinical bridges through a comprehensive therapy orientation, focus on stigma reduction, integration of cultural metaphors and symbols, and use of cultural and philosophical teachings.

The final evaluation of intervention efficacy will be conducted via a randomized controlled trial with 360 Asian American participants. Over 14 weeks (1 week for pretest + 12 weeks for intervention + 1 week for posttest), the investigators will assess whether, compared to a business-as-usual (BAU) or an active control (AC), implementation of the full PRoP-AA intervention: (a) increases social problem-solving, (b) increases participant self-efficacy, (c) decreases stress and depression, (d) increases motivation to engage with the intervention, (e) improves attitudes towards seeking mental health help, and (f) increases knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Chinese American
* ability to understand English, Mandarin, or Cantonese
* has access to a mobile device running Android or iOS

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Social problem-solving | Baseline and 12 weeks
  Social problem-solving will be measured using the Social Problem-Solving Inventory-Revised: Short Form (SPSI-R).The SPSI-R: Short Form is a 25-item multi-dimensional measure of social problem solving derived from a factor analysis of the original 70-item theory-driven Social Problem-Solving Inventory. In addition to a total score, it consists of five scales that measure two constructive dimensions (positive problem orientation, rational problem solving) and three dysfunctional dimensions (negative problem orientation, impulsivity/carelessness style, avoidance style).
Self-Efficacy | Baseline and 12 weeks
  Self-efficacy will be measured using the Mental Health Self-Efficacy Scale (MHSES), a 6-item Likert-type single-factor scale measuring one's capability to perform behaviors related to mental health. The MHSES has demonstrated good internal reliability (alpha = .89) and is positively correlated with work, social adjustment, and emotional stability, and negatively correlated with measures of depression.
Stress | Baseline and 12 weeks
  Stress will be assessed using the Depression Anxiety and Stress Scale-21 (DASS-21).128 The DAS-21 is a 21-item scale that measures three related negative states of depression, anxiety, and stress. It has shown strong internal reliability and moderate validity through confirmatory factor analysis,
Anxiety | Baseline and 12 weeks
  Anxiety will be assessed using the Depression Anxiety and Stress Scale-21 (DASS-21).128 The DAS-21 is a 21-item scale that measures three related negative states of depression, anxiety, and stress. It has shown strong internal reliability and moderate validity through confirmatory factor analysis,
Depression | Baseline and 12 weeks
  Depression will be assessed using the Depression Anxiety and Stress Scale-21 (DASS-21).128 The DAS-21 is a 21-item scale that measures three related negative states of depression, anxiety, and stress. It has shown strong internal reliability and moderate validity through confirmatory factor analysis,
Attitudes towards seeking mental help | Baseline and 12 weeks
  Attitudes towards seeking mental help will be assessed using the Mental Help Seeking Attitudes Scale (MHSAS) and the Perceived Devaluation and Discrimination Scale (PDD). The MHSAS a 9-item scale that measures participants' overall attitudes (positive or negative) towards seeking help from a mental health expert. The PDD is a 12-item scale that assesses stigma around mental health. Both the MHSAS and the PDD have demonstrated good internal consistency and test-retest reliability. The PDD has been used translated into Chinese.138 In addition to these two scales, the investigators will develop items to assess participants' attitudes towards using mHealth mental health applications specifically.
Knowledge | 12 weeks
  Knowledge will be measured using a multiple-choice survey that the project developed to determine the extent to which participants understand basic information delivered in the program around Problem-Solving Therapy skills and content.

SECONDARY OUTCOMES:
Loss of face | Baseline and 12 weeks
  Loss of face will be examined as a moderator of the effect of the program, and will be measured using the Loss of Face scale (LOF). The LOF is a 21-item, 7-point Likert-type scale that evaluates concern about violating social norms and concern about causing others to lose face. The LOF has demonstrated good internal reliability (alpha = .83), as well as concurrent and discriminant validity (correlating with other-directedness, private and public self-consciousness, and social anxiety).7 The LOF has been translated into Chinese.
Motivation to engage with the intervention | 12 weeks
  Motivation to engage with the intervention will be assessed using the Situational Motivation Scale (SIMS). The SIM is a 16-item Likert-type scale with four internally consistent factors (alphas > .77): intrinsic motivation, identified regulation, external regulation, and motivation. The SIMS has been used extensively to evaluate motivation in many contexts and towards many activities, including mandated training, and has been translated into Chinese.
Usability, content utility and validity, user satisfaction, and cultural relevance | 12 weeks
  Usability, content utility and validity, user satisfaction, and cultural relevance will be assessed with Likert-type scale items and open-ended questions. The investigators will measure the three evaluation areas for digital learning products: (1) interface usability (e.g., Was the application easy to use?), (2) content validity (e.g., Did the content make sense?), and (3) content utility (e.g., What did participants learn?). In addition to program-specific usability questions, the investigators will include the System Usability Scale (SUS) to assess overall usability, with minor wording changes to align the questions with the product being assessed and the addition of an adjective rating scale to help communicate the numeric results to those less familiar with usability studies.

CONTACTS AND LOCATIONS:
Locations (1):
- IrisEd dba Trifoia, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the final results of the project are accepted for publication all de-identified final research data and associated codebooks will be made accessible to interested researchers upon request to the PI and archived with the Inter-university Consortium for Political and Social Research (ICPSR).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the final report of the grant is submitted and associated publications are accepted we will make the de-identified final research data and associated codebooks available within 6 months.